CLINICAL TRIAL: NCT06716983
Title: Multimodal Investigation of Cortico-Basal Ganglia-Thalamo-Cortical (CBGTC) Network Dynamics in Dystonic Patients with Deep Brain Stimulation (DBS)
Brief Title: Multimodal Investigation of Cortico-Basal Ganglia-Thalamo-Cortical Network Dynamics in Dystonic Patients with Deep Brain Stimulation
Acronym: DYScover
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: DYScover; GR-2021-12375334 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-12-02; First posted 2024-12-04 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Dystonia
Keywords: Dystonia; Movement disorders; Deep Brain Stimulation; DBS; Local Field potentials; biomarker; Magnetoencephalography; MEG; fMRI
MeSH Terms: conditions — Dystonia; Movement Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples with DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: fMRI — fMRI in patients with dystonia implanted with deep brain stimulation with neurostimulators capable of recording local field potentials
Diagnostic Test: EEG-MEG — EEG-MEG in patients with dystonia implanted with deep brain stimulation with neurostimulators capable of recording local field potentials
Diagnostic Test: registration of local field potentials — registration of local field potential in patients with dystonia implanted with deep brain stimulation
Diagnostic Test: genetic panel — genetic panel for dystonia

SUMMARY:
The goal of this prospective open label study is to elucidate the pathophysiology of dystonia and to understand how deep brain stimulation (DBS) influences brain networks. The investigators will enroll patients with dystonia implanted with DBS of the Globus Pallidus internus (GPi) with sensing implantable neurostimulators, capable of measuring GPi local field potentials (LFPs).

The main questions it aims to answer are:

* does DBS influence pallidal LFPs in the long term?
* how the basal-ganglia-thalamo-cortical circuit is modified after DBS?
* do LFPs changes correlate with clinical improvement? Participants will undergo to serial clinical evaluations, magnetoencephalography (MEG) and functional Magnetic Resonance Imaging (fMRI) studies. Primarily, the data obtained from our study might help in clarifying basic pathological electrophysiological features of dystonia. These features might be secondarily used in future to provide a framework for an effective application of closed-loop DBS in Dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic or genetic dystonia who have already undergone DBS surgery of the globus pallidus internus
* Patient implanted with a neurostimulator capable of chronically recording LFPs and which is fully compatible with magnetic fields up to 3 Tesla.
* Age>12 years

Exclusion Criteria:

* Evidence of CNS pathology or any other acquired conditions (perinatal, infective, toxic, neoplastic, vascular, psychogenic) responsible for the dystonia phenomenology,
* Focal distribution of dystonia
* Contraindications to brain MRI or EEG/MEG
* Adult subjects unable to express consent to inclusion in the study
* Pregnancy, and breastfeeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will enroll 15 consecutive patients with idiopathic or genetic dystonia who have already undergone DBS surgery of the globus pallidus internus with a neurostimulator capable of chronically recording LFPs and which is fully compatible with magnetic fields up to 3 Tesla.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Local field potentials | 1 year
  To confirm the prominent pallidal low frequency oscillations in GPi (LFPs in alpha and theta bands) in dystonic patients and to evaluate the modifications in LFPs after DBS in the long term.

SECONDARY OUTCOMES:
Coherence LFPs-MEG | 1 year
  To evaluate coherence and/or correlation between GPi acivity and the neural activity in the basal ganglia-thalamo-cortical circuitry. LFPs signals will be co-registered to both EEG/MEG and resting state fMRI.
Clinical correlations | 1 year
  to find a correlation between modulation of pallidal low-frequency activity and patient's clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Levi, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

REFERENCES:
- [Background] Wang DD, de Hemptinne C, Miocinovic S, Ostrem JL, Galifianakis NB, San Luciano M, Starr PA. Pallidal Deep-Brain Stimulation Disrupts Pallidal Beta Oscillations and Coherence with Primary Motor Cortex in Parkinson's Disease. J Neurosci. 2018 May 9;38(19):4556-4568. doi: 10.1523/JNEUROSCI.0431-18.2018. Epub 2018 Apr 16. PMID 29661966
- [Background] Udupa K, Bhattacharya A, Chen R. Exploring the connections between basal ganglia and cortex revealed by transcranial magnetic stimulation, evoked potential and deep brain stimulation in dystonia. Eur J Paediatr Neurol. 2022 Jan;36:69-77. doi: 10.1016/j.ejpn.2021.12.004. Epub 2021 Dec 10. PMID 34922163
- [Background] Thenaisie Y, Palmisano C, Canessa A, Keulen BJ, Capetian P, Jimenez MC, Bally JF, Manferlotti E, Beccaria L, Zutt R, Courtine G, Bloch J, van der Gaag NA, Hoffmann CF, Moraud EM, Isaias IU, Contarino MF. Towards adaptive deep brain stimulation: clinical and technical notes on a novel commercial device for chronic brain sensing. J Neural Eng. 2021 Aug 31;18(4). doi: 10.1088/1741-2552/ac1d5b. PMID 34388744
- [Background] Talakoub O, Neagu B, Udupa K, Tsang E, Chen R, Popovic MR, Wong W. Time-course of coherence in the human basal ganglia during voluntary movements. Sci Rep. 2016 Oct 11;6:34930. doi: 10.1038/srep34930. PMID 27725721
- [Background] Sirica D, Hewitt AL, Tarolli CG, Weber MT, Zimmerman C, Santiago A, Wensel A, Mink JW, Lizarraga KJ. Neurophysiological biomarkers to optimize deep brain stimulation in movement disorders. Neurodegener Dis Manag. 2021 Aug;11(4):315-328. doi: 10.2217/nmt-2021-0002. Epub 2021 Jul 15. PMID 34261338
- [Background] Scheller U, Lofredi R, van Wijk BCM, Saryyeva A, Krauss JK, Schneider GH, Kroneberg D, Krause P, Neumann WJ, Kuhn AA. Pallidal low-frequency activity in dystonia after cessation of long-term deep brain stimulation. Mov Disord. 2019 Nov;34(11):1734-1739. doi: 10.1002/mds.27838. Epub 2019 Sep 4. PMID 31483903
- [Background] Prescott IA, Marino RA, Levy R. Field evoked potentials in the globus pallidus of non-human primates. Neurosci Res. 2017 Jul;120:18-27. doi: 10.1016/j.neures.2017.01.007. Epub 2017 Jan 31. PMID 28159649
- [Background] Pina-Fuentes D, Beudel M, Little S, van Zijl J, Elting JW, Oterdoom DLM, van Egmond ME, van Dijk JMC, Tijssen MAJ. Toward adaptive deep brain stimulation for dystonia. Neurosurg Focus. 2018 Aug;45(2):E3. doi: 10.3171/2018.5.FOCUS18155. PMID 30064317
- [Background] Neumann WJ, Jha A, Bock A, Huebl J, Horn A, Schneider GH, Sander TH, Litvak V, Kuhn AA. Cortico-pallidal oscillatory connectivity in patients with dystonia. Brain. 2015 Jul;138(Pt 7):1894-906. doi: 10.1093/brain/awv109. Epub 2015 May 1. PMID 25935723
- [Background] Litvak V, Florin E, Tamas G, Groppa S, Muthuraman M. EEG and MEG primers for tracking DBS network effects. Neuroimage. 2021 Jan 1;224:117447. doi: 10.1016/j.neuroimage.2020.117447. Epub 2020 Oct 12. PMID 33059051
- [Background] Harmsen IE, Rowland NC, Wennberg RA, Lozano AM. Characterizing the effects of deep brain stimulation with magnetoencephalography: A review. Brain Stimul. 2018 May-Jun;11(3):481-491. doi: 10.1016/j.brs.2017.12.016. Epub 2018 Jan 4. PMID 29331287
- [Background] Barow E, Neumann WJ, Brucke C, Huebl J, Horn A, Brown P, Krauss JK, Schneider GH, Kuhn AA. Deep brain stimulation suppresses pallidal low frequency activity in patients with phasic dystonic movements. Brain. 2014 Nov;137(Pt 11):3012-3024. doi: 10.1093/brain/awu258. Epub 2014 Sep 10. PMID 25212852
- [Background] Averna A, Arlotti M, Rosa M, Chabardes S, Seigneuret E, Priori A, Moro E, Meoni S. Pallidal and Cortical Oscillations in Freely Moving Patients With Dystonia. Neuromodulation. 2023 Dec;26(8):1661-1667. doi: 10.1111/ner.13503. Epub 2022 Feb 15. PMID 34328685